CLINICAL TRIAL: NCT02884375
Title: Elderly Cancer Patient: ELCAPA Cohort Survey
Brief Title: Elderly CAncer Patient
Acronym: ELCAPA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); Oncogeriatric Coordination Unit (UCOG) - Sud-Val-de-Marne (Unknown); Oncogeriatric Coordination Unit (UCOG) - Paris-Ouest (Unknown); Cancéropôle Ile De France (Unknown)
Responsible Party: Sponsor
Other Study IDs: UG 6729 UCOG
Record Dates: First submitted 2016-08-18; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Hematologic Malignancies; Solid Cancer
Keywords: Elderly; Cancer; Geriatric assessment; Treatment; Epidemiology
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly cancer patient cohort: Patients aged 70 years or older, who had diagnosis of cancer in participating sites (including hematologic malignancies), and referred to a geriatrician for geriatric assessment (GA)
  Interventions: Other: Extensive GA

INTERVENTIONS:
Other: Extensive GA — GA includes an evaluation of nine domains according to international recommendations :
  * functional status (six-item Activities of Daily Living (ADL) score, Instrumental Activities of Daily Living (IADL))
  * mobility (timed get-up-and-go test, one-leg standing balance test, history of fall)
  * nutritional status (French National Authority of Health guidelines, weight loss body mass index (BMI), Mini Nutritional Assessment, albumin )
  * cognitive status (Mini-Mental State Examination (MMSE), history of dementia, confusion)
  * mood (Mini-Geriatric Depression Scale (Mini-GDS), symptoms of anxiety, depression (DSM V))
  * comorbidities (CIRS G)
  * polypharmacy (number of medications)
  * social environment (primary caregiver, support at home, friends , family, living alone)
  * urinary and/or fecal incontinence

SUMMARY:
The management of older patients with cancer has become a major public health concern in Western countries because of the aging of the population and steady increase in cancer incidence with advancing age. Cancer treatment of aged patients is complex due to comorbidities, polypharmacy and functional status. The heterogeneity of the older population in terms of comorbidities and functional status may explain the difficulty in establishing management recommendations.

Study hypothesis is that a geriatric consultation using Geriatric Assessment (GA) can evaluate patient's resource and strengths, in order to help oncologist to define the most effective treatment. The GA developed by geriatricians and recommended by the International Society of Geriatric Oncology (SIOG), is a multidimensional assessment of general health status; comorbidities; functional status; nutritional, cognitive, psychological, and social parameters; and medications. The GA uses validated geriatric scales to produce an inventory of problems, which can then serve to develop an individualized geriatric intervention plan; it may be an important step in selecting elderly patients for cancer screening and treatment.

The objectives are:

* To assess the role of GA for decision making process for older patients with cancer
* To identify geriatric and oncologic factors associated with overall survival, treatment feasibility, toxicities, morbidities
* To develop and/or validate screening tests for frailty in geriatric oncology
* To develop and validate frailty classifications

Method: The ELCAPA (ELderly CAncer PAtient) survey is a French multicentric prospective study that includes all patients age 70 years or older who has a diagnosis of solid cancer or hematologic malignancies in French hospitals

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 70 years or older
* Diagnosed cancer at all stage
* Referred to a geriatrician for GA
* Given oral non-opposition from patient or a legally mandated person

Exclusion Criteria:

* Oral opposition

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients aged 70 years or older, who had diagnosis of cancer (including hematologic malignancies), and referred to a getrician for GA in participating sites
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-09; Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Difference between initial oncologist treatment proposal and final treatment selected after geriatric assessment | through multidisciplinary meeting decision, an average of 2 weeks after GA (+/-1 week).

SECONDARY OUTCOMES:
Chemotherapy toxicities using Common Terminology Criteria for Adverse Events | through chemotherapy treatment completion, an average of 6-months after inclusion (+/- 3 months) (according to curative or palliative and chemotherapy protocols).
Feasibility of the planned Chemotherapy treatment (delivery of the planned number of cycles determined based on tumor site and metastatic status) | through chemotherapy treatment completion, an average of 6-months after inclusion (+/- 3 months) (according to curative ou palliative and chemotherapy protocols).
Overall mortality | Year 1 and 5 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: PHILIPPE CAILLET, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; ELENA PAILLAUD, MD-PhD, Study Director — Assistance Publique - Hôpitaux de Paris; FLORENCE CANOUI-POITRINE, MD-PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Gonzalez Serrano A, Laurent M, Barnay T, Martinez-Tapia C, Audureau E, Boudou-Rouquette P, Aparicio T, Rollot-Trad F, Soubeyran P, Bellera C, Caillet P, Paillaud E, Canoui-Poitrine F. A Two-Step Frailty Assessment Strategy in Older Patients With Solid Tumors: A Decision Curve Analysis. J Clin Oncol. 2023 Feb 1;41(4):826-834. doi: 10.1200/JCO.22.01118. Epub 2022 Oct 28. PMID 36306481
- [Derived] Martinez-Tapia C, Diot T, Oubaya N, Paillaud E, Poisson J, Gisselbrecht M, Morisset L, Caillet P, Baudin A, Pamoukdjian F, Broussier A, Bastuji-Garin S, Laurent M, Canoui-Poitrine F. The obesity paradox for mid- and long-term mortality in older cancer patients: a prospective multicenter cohort study. Am J Clin Nutr. 2021 Jan;113(1):129-141. doi: 10.1093/ajcn/nqaa238. Epub 2020 Sep 5. PMID 32889525